CLINICAL TRIAL: NCT04105127
Title: Pain and Discomfort With Anterior Versus Posterior Builds-up During Fixed Orthodontic Treatment: a Randomized Clinical Trial
Brief Title: Pain and Discomfort With Anterior Versus Posterior Builds-up
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, ALESSANDRO UGOLINI, Assistant Professor, University of Genova
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT Builds-ups
Record Dates: First submitted 2019-06-06; First posted 2019-09-26 (Actual); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Malocclusion; Deep Bite
MeSH Terms: conditions — Malocclusion; Overbite

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Anterior builds-ups (Active Comparator): Intervention orthodontic - fixed orthodontic treatment in patients with overbite reduction: fixed orthodontic treatment with resin build-ups bonded to the palatal surfaces of central upper incisors
  Interventions: Device: orthodontic - Anterior resin builds-ups
- Posterior builds-ups (Active Comparator): Intervention orthodontic - fixed orthodontic treatment in patients with overbite reduction: fixed orthodontic treatment with resin build-ups bonded to the occlusal surfaces of first or second upper/lower molars
  Interventions: Device: orthodontic - Posterior resin builds-ups

INTERVENTIONS:
Device: orthodontic - Anterior resin builds-ups — After lower brackets placement, resin builds-ups are added on the palatal aspect of the upper central incisors. Both central incisors are customarily bonded to broadly distribute the occlusal forces. Builds-ups are removed when the overbite was considered adequate to prevent lower brackets detachment.
  Other Names: Anterior resin bite turbos
  Arms: Anterior builds-ups
Device: orthodontic - Posterior resin builds-ups — After lower brackets placement, resin builds-ups are added on the supporting cusps of first or second upper/lower molars. Builds-ups are removed when the overbite was considered adequate to prevent lower brackets detachment.
  Other Names: Posterior resin bite turbos
  Arms: Posterior builds-ups

SUMMARY:
Orthodontic build-ups are made by composite/resin material bonded to the palatal or occlusal surfaces of teeth (usually molars or incisors). Their primary purpose is to prevent heavy contact of the upper teeth with lower fixed appliances in patients with overbite reduction to avoid brackets detachment. These appliances disarticulate the posterior teeth, deprogram the masticatory muscles and allow for eruption, extrusion, and uprighting of the posterior teeth. Build-ups are usually placed in the first months of the fixed orthodontic treatment and contribute to increasing the perception of pain. In the orthodontic daily practice, the pain is the most frequent symptom during treatment and is the one that most frightens/worries the patients. Literature shows that fear of pain is one of the primary reasons that patients fail to seek orthodontic care. Pain has a negative effect on patients' compliance, oral hygiene, and missed appointments. Its effects on patients' daily lives is a major reason for discontinuance of orthodontic treatment.

In the literature the prevention of pain and management of orthodontic builds-ups is a poorly analyzed topic, despite being a daily problem in orthodontic clinical practice. So, the aim of the present study is to investigate and analyze the perception of pain and function impairment with different type of build-ups (anterior or posterior) to identify an efficient clinical management protocol and an effective pain and discomfort prevention strategy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with reduced overbite treated with orthodontic fixed appliance
* Angle Class I, Class II or Class III malocclusion

Exclusion Criteria:

* Hypodontia in any quadrant excluding third molars
* Craniofacial syndromes, or cleft lip or palate

Ages: 9 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2020-09-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Overbite correction [Millimeters] | 1 week
  Overbite Clinical evaluation in vivo (continuous outcome, millimeters)
Overbite correction [Millimeters] | 1 months
  Overbite Clinical evaluation in vivo (continuous outcome, millimeters)
Overbite correction [Millimeters] | 2 months
  Overbite Clinical evaluation in vivo (continuous outcome, millimeters)
Overbite correction [Millimeters] | 3 months
  Overbite Clinical evaluation in vivo (continuous outcome, millimeters)
Overbite correction [Time] | 1 months
  Overbite Clinical evaluation in vivo (continuous outcome, months)
Overbite correction [Time] | 2 months
  Overbite Clinical evaluation in vivo (continuous outcome, months)
Overbite correction [Time] | 3 months
  Overbite Clinical evaluation in vivo (continuous outcome, months)
Pain after builds-up placement | 1 week
  Visual Analogic Scale (VAS) were used to evaluate the level of pain. The Visual Analog Scale (VAS) is most commonly a straight 100-mm line, without demarcation, that has the words "no pain" at the left-most end and "worst pain imaginable" (or something similar) at the right-most end. Patients are instructed to place a mark on the line indicating the amount of pain that they feel at the time of the evaluation. The distance of this mark from the left end is then measured, and this number is used as a numeric representation of the severity of the patient's pain.
Pain after builds-up placement | 1 months
  Visual Analogic Scale (VAS) were used to evaluate the level of pain. The Visual Analog Scale (VAS) is most commonly a straight 100-mm line, without demarcation, that has the words "no pain" at the left-most end and "worst pain imaginable" (or something similar) at the right-most end. Patients are instructed to place a mark on the line indicating the amount of pain that they feel at the time of the evaluation. The distance of this mark from the left end is then measured, and this number is used as a numeric representation of the severity of the patient's pain.
Pain after builds-up placement | 2 months
  Visual Analogic Scale (VAS) were used to evaluate the level of pain. The Visual Analog Scale (VAS) is most commonly a straight 100-mm line, without demarcation, that has the words "no pain" at the left-most end and "worst pain imaginable" (or something similar) at the right-most end. Patients are instructed to place a mark on the line indicating the amount of pain that they feel at the time of the evaluation. The distance of this mark from the left end is then measured, and this number is used as a numeric representation of the severity of the patient's pain.
Pain after builds-up placement | 3 months
  Visual Analogic Scale (VAS) were used to evaluate the level of pain. The Visual Analog Scale (VAS) is most commonly a straight 100-mm line, without demarcation, that has the words "no pain" at the left-most end and "worst pain imaginable" (or something similar) at the right-most end. Patients are instructed to place a mark on the line indicating the amount of pain that they feel at the time of the evaluation. The distance of this mark from the left end is then measured, and this number is used as a numeric representation of the severity of the patient's pain.
Oral Health Impact Profile after builds-up placement | 1 week
  Instrument of data collection was OHIP-14 questionnaire, which comprises of 14 questions with two questions each under seven domains. The domains include; functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses to the questions are based on a Likert scale which ranged from 0- "never" to 4- "very often". Variables also included in the questionnaire were: demographic variables and satisfaction ratings of teeth appearance and self- rating of tooth condition. The satisfaction ratings of tooth appearance assessed how satisfied the participants were with the appearance of their teeth with a response of "satisfied or dissatisfied". The self- rating of tooth condition assessed oral condition as being "good or poor". The satisfaction ratings and self-ratings of oral health were variables used to assess the construct validity of OHIP-14 in the respondents
Oral Health Impact Profile after builds-up placement | 1 months
  Instrument of data collection was OHIP-14 questionnaire, which comprises of 14 questions with two questions each under seven domains. The domains include; functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses to the questions are based on a Likert scale which ranged from 0- "never" to 4- "very often". Variables also included in the questionnaire were: demographic variables and satisfaction ratings of teeth appearance and self- rating of tooth condition. The satisfaction ratings of tooth appearance assessed how satisfied the participants were with the appearance of their teeth with a response of "satisfied or dissatisfied". The self- rating of tooth condition assessed oral condition as being "good or poor". The satisfaction ratings and self-ratings of oral health were variables used to assess the construct validity of OHIP-14 in the respondents
Oral Health Impact Profile after builds-up placement | 2 months
  Instrument of data collection was OHIP-14 questionnaire, which comprises of 14 questions with two questions each under seven domains. The domains include; functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses to the questions are based on a Likert scale which ranged from 0- "never" to 4- "very often". Variables also included in the questionnaire were: demographic variables and satisfaction ratings of teeth appearance and self- rating of tooth condition. The satisfaction ratings of tooth appearance assessed how satisfied the participants were with the appearance of their teeth with a response of "satisfied or dissatisfied". The self- rating of tooth condition assessed oral condition as being "good or poor". The satisfaction ratings and self-ratings of oral health were variables used to assess the construct validity of OHIP-14 in the respondents
Oral Health Impact Profile after builds-up placement | 3 months
  Instrument of data collection was OHIP-14 questionnaire, which comprises of 14 questions with two questions each under seven domains. The domains include; functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability and handicap. Responses to the questions are based on a Likert scale which ranged from 0- "never" to 4- "very often". Variables also included in the questionnaire were: demographic variables and satisfaction ratings of teeth appearance and self- rating of tooth condition. The satisfaction ratings of tooth appearance assessed how satisfied the participants were with the appearance of their teeth with a response of "satisfied or dissatisfied". The self- rating of tooth condition assessed oral condition as being "good or poor". The satisfaction ratings and self-ratings of oral health were variables used to assess the construct validity of OHIP-14 in the respondents

CONTACTS AND LOCATIONS:
Locations (1):
- Alessandro Ugolini, Genova, GE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corridore D, Campus G, Guerra F, Ripari F, Sale S, Ottolenghi L. Validation of the Italian version of the Oral Health Impact Profile-14 (IOHIP-14). Ann Stomatol (Roma). 2014 Feb 4;4(3-4):239-43. eCollection 2013 Jul-Dec. PMID 24611088
- [Result] Kravitz ND, Jorgensen G, Frey S, Cope J. Resin bite turbos. J Clin Orthod. 2018 Sep;52(9):456-461. No abstract available. PMID 30256220
- [Result] Antoun JS, Thomson WM, Merriman TR, Rongo R, Farella M. Impact of skeletal divergence on oral health-related quality of life and self-reported jaw function. Korean J Orthod. 2017 May;47(3):186-194. doi: 10.4041/kjod.2017.47.3.186. Epub 2017 Mar 13. PMID 28523245
- [Result] Pativetpinyo D, Supronsinchai W, Changsiripun C. Immediate effects of temporary bite-raising with light-cured orthodontic band cement on the electromyographic response of masticatory muscles. J Appl Oral Sci. 2018 May 14;26:e20170214. doi: 10.1590/1678-7757-2017-0214. PMID 29768521